CLINICAL TRIAL: NCT06659575
Title: Prevalence of Sleep Disturbances in Elderly People Hospitalized in Medicine, Psychiatry and Rehabilitation Departments: TOPASE Prospective Study, RIPH 3
Acronym: TOPASE
Status: Completed | Type: Observational
Sponsor: University Hospital, Angers (Other Government)
Responsible Party: Sponsor
Other Study IDs: 49RC24_0305; 2024-A01996-41 (Other: ANSM)
Record Dates: First submitted 2024-10-14; First posted 2024-10-26 (Actual); Last update posted 2025-08-28 (Actual); Status verified 2025-08

CONDITIONS: D012893; Sleep Disorder
Keywords: Sleep Wake Disorders; Sleep; elderly; hospitalized; recovery process; rehospitalizations; overmedication; iatrogenics; daytime sleepiness; fatigue
MeSH Terms: conditions — Sleep Wake Disorders; Disorders of Excessive Somnolence; Fatigue

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients aged 60 and over hospitalized, expected length of stay > 48 hours: Inclusion criteria
  * Patients aged 60 and over hospitalized in a conventional medicine, psychiatry or medical and rehabilitation department of one of the GHT 49 healthcare establishments,
  * expected length of stay > 48 hours.
  Non-inclusion criteria
  * Patient hospitalized for more than 24 hours,
  * Inability to answer a questionnaire (assessment by the investigator or the medical team in charge of the patient (dementia, etc.),
  * No command of French,
  * Patient hospitalized for sleep pathology (evaluation or treatment),
  * Patient hospitalized in an intensive psychiatric care room,
  * Patients hospitalized under duress,
  * Patient opposition,
  * Patient under guardianship or curatorship.

SUMMARY:
Objectives and evaluation criteria:

The main objective of this study is to evaluate changes in sleep quality in patients aged 60 and over since their admission to a medical, psychiatric or medical and rehabilitation ward in one of the GHT 49 healthcare establishments.

The primary endpoint will be the difference between the usual sleep quality score and the sleep quality score during hospitalization, according to the Spiegel scale.

Research plan and procedure:

Patients participating in the study will be asked to complete a questionnaire including the Spiegel scale at two points during their hospitalization:

* Day 0: questionnaire n°1 to assess sleep quality on the night prior to hospitalization, including the Spiegel scale.
* Day 2 (morning of the third day of hospitalization): during the morning, depending on the organization of the ward, questionnaire n°2 to assess sleep quality during the previous night, including the Spiegel scale.

Number of research participants:

As the study is essentially descriptive, aimed at taking stock of the situation, the calculation of the number of patients to be included was not based on a hypothesis test.

Pragmatically, the investigator plan to include the maximum number of patients meeting the criteria during the targeted week.

Given the number of beds in the GHT 49 establishments in the departments concerned, and the average number of new admissions, the investigator estimate that 200 patients could be included.

Research duration:

Inclusion period: 5 days, Monday to Friday Participation period: 3 days (from day 0 to day 2) Study duration: 7 days

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 60 and over hospitalized in a conventional medicine, psychiatry or medical and rehabilitation department of one of the GHT 49 healthcare establishments,
* Anticipated hospital stay > 48 hours

Exclusion Criteria:

* Patient hospitalized for more than 24 hours,
* Inability to answer a questionnaire (assessment by the investigator or the medical team in charge of the patient (dementia, etc.),
* No mastery of French
* Patient hospitalized for sleep pathology (evaluation or treatment),
* Patient hospitalized in an intensive psychiatric care room,
* Patients hospitalized under duress,
* Patient opposition,
* Patient under guardianship or curatorship.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: As the study is essentially descriptive, aimed at taking stock of the situation, the calculation of the number of patients to be included was not based on a hypothesis test.
  Pragmatically, the investigator plan to include the maximum number of patients meeting the criteria during the targeted week.
  Given the number of beds in the GHT 49 establishments in the departments concerned, and the average number of new admissions, the investigator estimate that 200 patients could be included.
Sampling Method: Non-Probability Sample
Enrollment: 104 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-01-26 (Actual); Study Completion 2025-01-26 (Actual)

PRIMARY OUTCOMES:
The difference between the usual sleep quality score and the sleep quality score during hospitalization, according to the Spiegel scale. | 3 days
  The main objective of this study is to evaluate changes in sleep quality in patients aged 60 and over since their admission to a medical, psychiatric or medical and rehabilitation ward in one of the GHT 49 healthcare establishments.
  The primary endpoint will be the difference between the usual sleep quality score and the sleep quality score during hospitalization, according to the Spiegel scale.
  Patients participating in the study will be asked to complete a questionnaire including the Spiegel scale at two points during their hospitalization:
  * Day 0: questionnaire n°1 to assess sleep quality on the night prior to hospitalization, including the Spiegel scale.
  * Day 2 (morning of the third day of hospitalization): during the morning, depending on the organization of the ward, questionnaire n°2 to assess sleep quality during the previous night, including the Spiegel scale.
  NB: - Spiegel score ranks from 0 to 30 (Questionnaire)

SECONDARY OUTCOMES:
Participants numbers repartitions within departments categories following their spiegel score | 3 days
  * There is three categories: conventional medicine, psychiatry or medical care and rehabilitation.
  * Spiegel score ranks from 0 to 30 (Questionnaire)
Distributions of the number of participants within hospital facility types following their Spiegel score | 3 days
  * Four hospital categories: university hospitals, city hospitals, specialized hospitals and community hospitasl.
  * Spiegel score ranks from 0 to 30
Distribution of the number of participants in the different room types according to their Spiegel score | 3 days
  * Three different room types: Single or double without roomate and full double room
  * Spiegel score ranks from 0 to 30
Distributions of the number of participants by age group following Spiegel score | 3 days
  * Three age categories: 60-74 years, 75-89 years, 90 years and above
  * Spiegel score ranks from 0 to 30
Distribution of number of participants by gender and Spiegel score | 3 days
  * Gender
  * Spiegel score ranks from 0 to 30
Distribution of the number of patients within a list of different reported causes of sleep disorders (Questionnaire). | 3 days
  Was your sleep disturbed last night? 0 No 1 Yes
  If yes :
  * Anxiety
  * Need to go to the toilet
  * Noise
  * Change in rhythm of life (mealtimes, bedtimes, toilet times, etc.)
  * Medical devices (e.g. infusion, urinary catheter, dressing, etc.)
  * Pain
  * Light
  * My illness (clinical signs)
  * Lack of physical activity during the day
  * Smell
  * Visits from carers
  * Taking medication to sleep / absence / modification of usual treatment
  * Quality of bedding
  * Feeling hungry or thirsty
  * Room temperature
  * Room neighbor
  * Other : ________________________________________________

CONTACTS AND LOCATIONS:
Locations (10):
- France (10):
  - Angers_CHU, Angers
  - Etablissement de santé Baugeois-Vallée, Baugé-en-Anjou
  - CH de la corniche angevine, Chalonnes-sur-Loire
  - Cholet_Ch, Cholet
  - CH intercommunal Lys-Hyrôme, Cholet
  - Césame, Sainte-Gemmes-sur-Loire
  - CH Longué-Jumelles, Saumur
  - Saumur_Ch, Saumur
  - CH Doué-en-Anjou, Saumur
  - CH Layon-Aubance, Thouarcé

IPD SHARING:
Plan to Share IPD: Undecided